CLINICAL TRIAL: NCT01510652
Title: More Options Available With a Quadripolar Left Ventricular (LV) Lead pRovidE In-clinic Solutions to Cardiac Resynchronization Therapy (CRT) Challenges
Brief Title: More Options Available With a Quadripolar LV Lead pRovidE In-clinic Solutions to CRT Challenges
Acronym: MORE-CRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-11-006-HF-ID
Record Dates: First submitted 2011-11-30; First posted 2012-01-16 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Postoperative Cardiac Complication; Heart Failure; Left Ventricular Cardiac Dysfunction; Inappropriate Phrenic Nerve Stimulation; Perioperative/Postoperative Complications
Keywords: Cardiac Resynchronization therapy,; Heart Failure,; Left Ventricular Lead,; Quadripolar Left ventricular Lead,; Phrenic Nerve Stimulation,; Intra and post operative related complications
MeSH Terms: conditions — Heart Failure; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quad Group (Active Comparator): Patients in the Quad group will be implanted with St. Jude Medical (SJM) quadripolar Left Ventricular (LV) lead Quartet
  Interventions: Device: Quad Group
- BiP Group (Active Comparator): Patients in the BiP Group will be implanted with a standard (regulatory approved and commercially available) bipolar left ventricular lead from other companies (non St. Jude Medical leads)
  Interventions: Procedure: BiP Group

INTERVENTIONS:
Procedure: BiP Group — Implantation of standard Left Ventricular (LV) lead
  Arms: BiP Group
Device: Quad Group — Implantation of quadripolar Left ventricular (LV) lead Quartet
  Arms: Quad Group

SUMMARY:
This investigation is designed with the hypothesis that using a quadripolar left ventricular lead results in less interventions when dealing with high pacing thresholds and Phrenic Nerve Stimulation (PNS), both at implant and during follow-up, compared to standard bipolar left ventricular leads.

ELIGIBILITY:
Inclusion Criteria:

* Patients are indicated for Cardiac Resynchronization Therapy with Defibrillation backup device (CRT-D) implantation, as per current international certified guidelines
* Patients age is 18 years or greater
* Patients must indicate their understanding of the study and willingness to participate by signing the appropriate informed consent form
* Patients must be willing and able to comply with all study requirements

Exclusion Criteria:

* Patients with a life expectancy <12 months.
* Patients who are or may potentially be pregnant.
* Patient has suffered any of the following in the 4 weeks prior to enrolment:

  * Myocardial Infarction (MI)
  * Coronary Artery Bypass Graft (CABG)
  * Unstable Angina Pectoris
* Patient has primary valvular disease which has not been corrected

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1078 (Actual)
Dates: Start 2011-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Boriani, Pro., Principal Investigator — Policlinico Universitario S. Orsola e Malpighi, Bologna, Italy
Locations (64):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Hopital La Citadelle, Liège
- Canada (5):
  - Foothills Medical Center, Calgary
  - Royal Alexandra Hospital, Edmonton
  - QE II Health Sciences, Halifax
  - Institut de Cardiologie du Quebec - Hopital Laval, Québec
  - HSC Heastern Health, St. Johns
- Finland (2):
  - Paijat-Hame Central Hospital, Lahti
  - Tampere University Hospital, Tampere
- France (12):
  - CHU La Cavale Blanche, Brest
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHRU Hopital Albert Michallon, Grenoble
  - Hopital Cardiovasculaire et Pneumologique Louis Pradel, Lyon
  - Hopital de la Timone, Marseille
  - Hopital du Nord - CH Bourrely St. Antoine, Marseille
  - CHU Hopital G&R Laennec, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHRU Hopital de Pontchaillou, Rennes
  - CHRU Hopital Charles Nicolle, Rouen
  - CHU St. Etienne, Saint-Priest-en-Jarez
  - Clinique du Tonkin, Villeurbanne
- Germany (11):
  - Charite Campus Virchow Klinikum, Berlin
  - Unfallkrankenhaus Berlin-Marzahn, Berlin
  - Stadtische Kliniken Bielefeld, Bielefeld
  - Klinikum Coburg, Coburg
  - Elisabeth-Krankenhaus, Essen
  - Universitatsklinikum Greifswald, Greifswald
  - Universitatskliniken des Saarlandes, Homburg
  - Universitatsklinikum Leipzig, Leipzig
  - Stadtisches Klinikum Ludwigshafen, Ludwigshafen
  - Klinikum Ludenscheid, Lüdenscheid
  - Krankenhaus der Barmherzigen, Trier
- India (2):
  - All India Institute of Medical Sciences, New Delhi
  - Escorts Heart Institute and Research Center, New Delhi
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Soroka University Hospital, Beersheba
  - Kaplan Medical Center, Rehovot
  - Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Policlinico S. Orsola & Malpighi, Bologna
  - Azienda Ospedaliera S.Anna e S.Sebastiano, Caserta
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Ospedale Vito Fazzi, Lecce
  - Ospedale Maggiore della Carità, Novara
  - Policlinico Casilino, Rome
  - Ospedale SS. Annunziata, Taranto
  - Azienda Sanitaria Ospedaliera Molinette S. Giovanni Battista, Torino
  - Ospedale Civile Maggiore Verona Borgo Trento, Verona
- Netherlands (4):
  - Amphia Hospital, Breda
  - Medisch Spectrum Twente, Enschede
  - Haga Ziekenhuis, The Hague
  - MC Haaglanden, The Hague
- Slaskie Centrum Chorob Serca, Zabrze, Poland
- Spain (3):
  - Hospital de Basurto, Bilbao
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitari La Fe, Valencia
- Switzerland (4):
  - Basel University Hospital, Basel
  - Hopital Cantonal Universitaire de Geneva, Geneva
  - Fondazione Cardiocentro Ticino, Lugano
  - Universitaets Spital Zuerich, Zurich
- United Kingdom (5):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Bournemouth Hospital, Bournemouth
  - University Hospital of Wales, Cardiff
  - St. Thomas Hospital, London
  - James Cook University Hospital, Middlesbrough

REFERENCES:
- [Derived] Boriani G, Connors S, Kalarus Z, Lemke B, Mullens W, Osca Asensi J, Raatikainen P, Gazzola C, Farazi TG, Leclercq C. Cardiac Resynchronization Therapy With a Quadripolar Electrode Lead Decreases Complications at 6 Months: Results of the MORE-CRT Randomized Trial. JACC Clin Electrophysiol. 2016 Apr;2(2):212-220. doi: 10.1016/j.jacep.2015.10.004. Epub 2015 Nov 11. PMID 29766873

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1078 patients have been enrolled in this study, while 1074 have been randomized to Quad or BiP group.
  The randomization procedure happened after the enrollment and before the implant, this explains why not all 1078 patients have been randomized
Groups:
- Quad Group: Patients in the Quad group will be implanted with St. Jude Medical (SJM) quadripolar Left Ventricular (LV) lead Quartet
  Quartet Left Ventricular (LV) lead: Implantation of quadripolar Left ventricular (LV) lead Quartet
- BiP Group: Patients in the BiP Group will be implanted with a standard (regulatory approved and commercially available) bipolar left ventricular lead from other companies (non St. Jude Medical leads)
  Standard Left Ventricular (LV) lead: Implantation of standard Left Ventricular (LV) lead
Period: Overall Study
Arm/Group | Quad Group | BiP Group
Started | 719 | 355
Baseline | 718 | 348
Completed | 627 | 288
Not Completed | 92 | 67

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Quad Group | BiP Group | Total
Number analyzed (Participants) | 718 | 348 | 1066
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (10.2) | 68.4 (9.7) | 67.9 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 74 | 247
  Male | 545 | 274 | 819
Left Ventricular Ejection Fraction (LVEF) [Mean (Standard Deviation); unit: %] | 27.1 (7.6) | 27.5 (8.1) | 27.2 (7.7)
Left Ventricular End-Diastolic Volume (LVEDV) [Mean (Standard Deviation); unit: ml] | 200.4 (74.9) | 204.5 (72.0) | 203.2 (80.6)
Left Ventricular End-Systolic Volume (LVESV) [Mean (Standard Deviation); unit: ml] | 151.2 (64.0) | 149.0 (58.3) | 150.5 (62.2)
QRS duration [Mean (Standard Deviation); unit: ms] | 158 (29) | 157 (27) | 157.5 (28.4)
Cardiomyopathy [Number; unit: participants]
  Ischemic | 353 | 196 | 549
  Non Ischemic | 365 | 152 | 517
Atrial Arrhythmia History [Number; unit: participants]
  Atrial Fibrillation | 114 | 58 | 172
  Atrial Flutter | 21 | 7 | 28
  None | 583 | 283 | 866

OUTCOME MEASURES:

1. Primary Outcome: Lead Performance
Description: Percentage of patients with freedom from event (intra- and post-operative). Intra-operative events were defined as: need to use more than 1 left ventricular lead, need to change lead implant position, use of any device to actively fixate the lead, unsuccessful implant, due to phrenic nerve stimulation, high pacing threshold or lead instability.
  Post-operative events were defined as any left ventricular lead related serious adverse device effect and CRT switched off.
Time Frame: 6 months
Measure: Number; unit: % of patients with freedom from event
Arm/Group | Quad Group | BiP Group
Number analyzed (Participants) | 719 | 355
% of patients with freedom from event | 83 | 74.4

2. Secondary Outcome: Percentage of Cardiac Resynchronization Therapy Responders
Description: Percentage of Cardiac Resynchronization Therapy (CRT) responders measured by a decrease of at least 10% of Left Ventricle End-Systolic Volume (LVESV)
Time Frame: Baseline and 6 months
Population: The number of participants analyzed is the number of patients with echo data received for both baseline and 6 months follow up visits (and so comparable)
Measure: Number; unit: % of patients that are CRT responders
Arm/Group | Quad Group | BiP Group
Number analyzed (Participants) | 476 | 218
% of patients that are CRT responders | 62.0 | 56.0

3. Secondary Outcome: Implant Duration
Description: This measure reports the length (in time) of the implantation procedure. The measurement start at skin incision and stop at skin suture (so called skin-to-skin time) The total implant procedure duration time will be compared between the control and the treatment group.
Time Frame: Total duration of the implant procedure reported at the end of the procedure
Population: The number of participants analyzed is the number of patients with implant data duration time available.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Quad Group | BiP Group
Number analyzed (Participants) | 710 | 342
min | 100.4 (54.5) | 101.1 (51)

ADVERSE EVENTS:
Time Frame: 6 Months: From the enrollment to 6 Months Follow Up
Arm/Group | Quad Group | BiP Group
Serious Adverse Events (participants affected / at risk) | 332/719 | 211/355
Other Adverse Events (participants affected / at risk) | 186/719 | 76/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad Group (N=719) | BiP Group (N=355)
Arrhythmia (Cardiac disorders) | 53 (55) | 35 (35)
Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Heart Failure (Cardiac disorders) | 41 (55) | 24 (30)
Hematoma (Injury, poisoning and procedural complications) | 16 (16) | 9 (9)
Infection (Infections and infestations) | 24 (24) | 22 (22)
Lead Dislodgement (LV Lead) (Surgical and medical procedures) | 37 (37) | 20 (22)
Lead Fracture (LV Lead) (Surgical and medical procedures) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Phrenic Nerve Stimulation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (8)
Other - Non Cardiac (General disorders) | 81 (83) | 48 (51)
Other - Cardiac (Cardiac disorders) | 20 (21) | 9 (9)
Cardiac Perforation (RV Lead) (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Cardiac Tamponade (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Coronary Sinus Dissection (LV Lead related) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Death for Unknown Causes (General disorders) | 5 (5) | 3 (3)
Pocket Erosion (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 2 (2) | 2 (2)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Coronary Sinus Dissection (Other Device related) (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lead Dislodgement (RA Lead) (Surgical and medical procedures) | 7 (9) | 5 (5)
Lead Dislodgement (RV Lead) (Surgical and medical procedures) | 15 (15) | 5 (5)
Lead Fracture (RV Lead) (Surgical and medical procedures) | 1 (2) | 0 (0)
Lead Malfunction (RA Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)
Lead Unstable Position (LV Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)
Loss of Capture (RV Lead) (Surgical and medical procedures) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quad Group (N=719) | BiP Group (N=355)
Arrhythmia (Cardiac disorders) | 28 (29) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 4 (6)
Heart Failure (Cardiac disorders) | 8 (8) | 10 (10)
Hematoma (Injury, poisoning and procedural complications) | 25 (25) | 6 (8)
Infection (Infections and infestations) | 6 (6) | 2 (2)
Lead Damaged during Implant (Surgical and medical procedures) | 1 (1) | 0 (0)
Lead Dislodgement (LV Lead) (Surgical and medical procedures) | 7 (7) | 3 (3)
Phrenic Nerve stimulation (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 11 (14)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Other - Non Cardiac (General disorders) | 42 (43) | 16 (16)
Cardiac Perforation (Other Device Related) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Other - Cardiac (Cardiac disorders) | 19 (24) | 12 (12)
Coronary Sinus Dissection (LV Lead Related) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Coronary Sinus Dissection (Other Device Related) (Surgical and medical procedures) | 6 (6) | 2 (2)
High Voltage Lead Impedance (RV Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)
Lead Dislodgement (RA Lead) (Surgical and medical procedures) | 1 (1) | 1 (1)
Loss Of Capture (LV Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)
Oversensing (RV Lead) (Surgical and medical procedures) | 2 (2) | 0 (0)
Pacing Impedance Out Of Range (LV Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)
Pacing Impedance Out Of Range (RV Lead) (Surgical and medical procedures) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Patients were followed for only 6 months, studies with longer follow-up would add to the body of evidence.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less